CLINICAL TRIAL: NCT00251082
Title: A Randomized, Placebo-Controlled, Double-Blind, Multi-National Study to Demonstrate Efficacy of Continuous Combined 0.5 mg Estradiol and 2.5 mg Dydrogesterone in the Treatment of Vasomotor Symptoms in Postmenopausal Women in Comparison to Placebo Over 3 Months, and to Investigate the Bleeding Pattern Over a Double-Blind Treatment Period of One Year Compared With Continuous Combined 1 mg Estradiol and 5 mg Dydrogesterone
Brief Title: Vasomotoric Symptoms Study of a 0.5 mg Estradiol and 2.5 mg Dydrogesterone Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Gregor Eibes, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S102.3.119; 2004-00215-25
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Postmenopause
Keywords: hormone replacement; vasomotoric symptoms; bleeding pattern
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: continuous combined estradiol and dydrogesterone
- B (Active Comparator)
  Interventions: Drug: continuous combined estradiol and dydrogesterone
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: continuous combined estradiol and dydrogesterone — 0.5 Mg Estradiol and 2.5 Mg Dydrogesterone
  Arms: A
Drug: continuous combined estradiol and dydrogesterone — 1 Mg Estradiol and 5 Mg Dydrogesterone
  Arms: B
Drug: Placebo — Placebo
  Arms: C

SUMMARY:
To demonstrate efficacy of continuous combined 0.5 mg estradiol and 2.5 mg dydrogesterone versus placebo in the treatment of vasomotor symptoms after a treatment period of 3 months and to investigate the bleeding pattern over a treatment period of one year

ELIGIBILITY:
Inclusion Criteria:

* Non-hysterectomised postmenopausal women
* Amenorrhoea for >= 12 months
* Serum estradiol and follicle stimulating hormone (FSH) in the postmenopausal range

Exclusion Criteria:

* Known hypersensitivity to estradiol, dydrogesterone or any of the excipients of the study medication
* Baseline endometrial biopsy result other than described in the inclusion criteria (no endometrial tissue for diagnosis, hyperplasia, carcinoma).
* Insufficient endometrial tissue for diagnosis obtained at baseline biopsy and endometrial thickness >= 5 mm (double layer) by transvaginal ultrasound.
* The presence of an endometrial polyp at baseline.
* Abnormal (un-investigated and/or unexplained) vaginal bleeding in the last 12 months prior to Screening Visit (Visit 1).
* Estradiol pellet/implant therapy during the past 6 months.
* Previous systemic unopposed estrogen replacement therapy over 6 months or more.
* History or presence of malignant neoplasms other than basal or spinal cell carcinoma of the skin

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The change in the number of moderate to severe hot flushes from baseline to week 13 | 12 weeks

SECONDARY OUTCOMES:
Change in the number of hot flushes from baseline to week 13; Change in the number of hot flushes and moderate to severe hot flushes from baseline to weeks 4 and 8; | 12 weeks
Change in the Menopause Rating Scale from baseline to weeks 4 and 13; | 52 weeks
Number of days with bleeding/spotting; Number of bleeding/spotting episodes; Number of days with a certain bleeding intensity (e.g. bleeding intensity =2); | 52 weeks
Length of bleeding free intervals; Amenorrhoea yes/no (absence of spotting and bleeding); Absence of bleeding yes/no; | 52 weeks
QualiPause Inventory 7D: weighted sum score of the symptoms | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (18):
- Croatia (3):
  - Site 11, Zagreb
  - Site 12, Zagreb
  - Site 13, Zagreb
- France (4):
  - Site 23, Cannes
  - Site 24, Cannes
  - Site 21, Montpellier
  - Site 22, Montpellier
- Poland (4):
  - Site 34, Katowice
  - Site 33, Krakow
  - Site 32, Lódź
  - Site 31, Warsaw
- Romania (4):
  - Site 41, Bucharest
  - Site 42, Bucharest
  - Site 44, Bucharest
  - Site 43, Craiova, Jud.Dolj
- Russia (3):
  - Site 51, Moscow
  - Site 52, Moscow
  - Site 53, Moscow